CLINICAL TRIAL: NCT07258537
Title: Modified Sims Versus Lumbar Roll Manipulation in Patients With Sacroiliac Joint Dysfunction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPTH02193002
Record Dates: First submitted 2025-07-22; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): modified SIM
  Interventions: Other: modified SIM manipulation

INTERVENTIONS:
Other: modified SIM manipulation — manipulation

SUMMARY:
This randomized controlled trial aims to compare the efficacy of two manual therapy techniques. Modified Sims Manipulation and Lumbar Roll Manipulation in treating Sacroiliac Joint Dysfunction (SIJD). The study will examine their effects on pain, quality of life, and well-being.

DETAILED DESCRIPTION:
The study investigates the short- and long-term therapeutic benefits of two different high-velocity low-amplitude thrust techniques, specifically Modified Sims and Lumbar Roll Manipulation, administered along with conventional therapy. Outcomes will be measured using NPRS, SF-36, WHO-5, and gait analysis (MaxTRAQ). Patients will be randomly assigned and blinded to the treatment group. Data collection will be conducted at Rasool Medical Complex, Gujrat.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-50

Either gender

Chronic LBP >1 month

3 or more positive SIJ provocation/motion tests

NPRS ≥3 at baseline

Exclusion Criteria:

Pelvic fracture

MRI-confirmed nerve root compression

Psoriatic/Reactive Arthritis

Elevated ESR/CRP

Neurological signs

Severe pain (NPRS >8)

Other red flags (malignancy, fever, etc.)

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale | 6 weeks
  Numeric pain rating scale: ranging from 0 ("no pain") to 10 ("worst possible pain")

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ashfaq Ahmed, PHD PT, Study Director — University of Lahore
Locations (1):
- Rasool Medical Complex, Gujrat, Punjab Province, Pakistan